CLINICAL TRIAL: NCT03710369
Title: Ergogenic Effect of PDE-5 Inhibitors at Moderate Altitude
Brief Title: Endurance Performance at Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Michael Koehle, Dr. Michael Koehle, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: H14-01736
Record Dates: First submitted 2015-11-23; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Altitude; Hypoxia; Sildenafil; Exercise
MeSH Terms: conditions — Hypoxia; Motor Activity | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Normoxia (Sham Comparator): Exercise in room air (normoxia). Sildenafil
  Interventions: Drug: Sildenafil
- Hypoxia (Active Comparator): Exercise in hypoxic air (reduced O2 concentration) that simulates 2500m elevation for 30-40 minutes with Sildenafil. Placebo
  Interventions: Drug: Placebo; Drug: Sildenafil

INTERVENTIONS:
Drug: Placebo — The placebo pill was compounded by McDonalds Pharmacy.
  Other Names: McDonalds Pharmacy
  Arms: Hypoxia
Drug: Sildenafil — Sildenafil from Pfizer, compounded by McDonalds Pharmacy.
  Other Names: Pfizer

SUMMARY:
The degree to which endurance exercise performance is diminished in acute hypoxia is variable and appears to be the result of several different physiological processes, however this research focuses on hypoxic pulmonary vasoconstriction (HPV). Sildenafil, a pulmonary vasodilator, has been used with mixed results to improve athletic performance in hypoxia. Because sildenafil has been shown to reduce HPV in some individuals, we believe that its effectiveness is closely related to the magnitude of the HPV response and the degree that individual exercise performance declines in hypoxia. This research will investigate the relationship between sildenafil, HPV, and exercise performance.

DETAILED DESCRIPTION:
1. Purpose

   The purpose of this research proposal is to evaluate the role of hypoxic pulmonary vasoconstriction (HPV) and the formation of arteriovenous anastomoses (shunts) in hypoxia and their effect on endurance exercise performance. The pulmonary vasodilator sildenafil will be used to reverse the effects of HPV during exercise. Large between-subject variability in exercise performance in hypoxia could be explained by similar variability in the HPV response. Elite and recreational athletes could benefit significantly from being aware of their HPV response to hypoxia and could alter their training accordingly based on this knowledge. The vasodilator sildenafil may provide a level playing field for those athletes who are compromised by a robust HPV response.
2. Hypothesis

   A greater decline in exercise performance in acute moderate hypoxia (FIO2 = 0.16) will be correlated with a higher pulmonary artery pressure (PAP) during steady-state exercise and resting in hypoxia, increased arteriovenous anastomoses in hypoxia, and a lower hypoxic ventilatory response (HVR). These subjects will have significantly improved exercise performance in hypoxia with sildenafil administration. This increase in performance will be associated with reduced PAP and increases in cardiac output.
3. Justification

   Professional athletic competitions are frequently held at moderate altitude: 1500-2999 meters, or a barometric pressure (PB) of 635-525 mmHg. These competitions include sports such as sky-running competitions and ski randonnée racing as well as Olympic competitions, for example the 1968 Mexico City Olympics, held at an altitude of 2,240 meters.

   Reasons for holding a competition at altitude vary. Some event host cities have venues that are situated at moderate altitude. Winter events that require a significant snowpack, such as Nordic and alpine ski races, are routinely held above 1500 meters. Finally, some athletes such as track cyclists and long track speed skaters may seek out moderate altitude venues where decreased atmospheric pressure reduces aerodynamic drag.

   As elevation increases above sea level, PB decreases. While the fractional concentration remains the same, this decrease reduces the partial pressures of the individual gases that make up the ambient air (primarily: oxygen, nitrogen, carbon dioxide). Decreased PB causes a reduction in the partial pressure of oxygen (PO2), resulting in less oxygen per given volume of air (hypoxia). The effects of reduced PB and the resultant physiologic effects of hypoxia on athletes are significant.

   The human respiratory system responds to hypoxia with hypoxic pulmonary vasoconstriction. In the lung, each alveolus is surrounded by a mesh-like network of blood vessels (capillaries). An important concern in respiratory physiology is the matching of blood flow to pulmonary ventilation, called the ventilation-perfusion (V/Q) ratio. When V/Q mismatch occurs, oxygen transport from the airspace of the lung to the tissues is disrupted. The HPV response acts to improve V/Q mismatch in hypoxia by directing blood flow away from under-ventilated (hypoxic) lung units and towards lung units that are receiving adequate ventilation. This is a useful response in the case of local hypoxia, for example, if a patient inhales a foreign object that becomes lodged in a bronchiole in the lung, airflow to the downstream lung units is impeded. The HPV response directs blood flow away from the hypoxic lung units and towards the other, better-ventilated parts of the lung where it can be properly oxygenated. This change in blood flow occurs at the pre-capillary level where smooth muscles surrounding the pulmonary arterioles constrict to close the vessels. This example of the HPV response to local hypoxia is beneficial to overall gas exchange. In the case of global hypoxia, at altitude, the HPV response may not be helpful and may in fact reduce oxygen transport. In global hypoxia, where all lung units are hypoxic, the HPV response still occurs, reducing blood flow throughout the lung even though the ideal response would be a global increase in blood flow to maximise the ability to transport O2.

   The result of the HPV response in global hypoxia is a marked increase in the pressure of the pulmonary artery (PAP), further increased during moderate and intense exercise. Increases in PAP lead to decreased stroke volume and cardiac output (Q). Because Qmax cannot increase, at any given workload Q is a higher fraction of Qmax. When exercising maximally, VO2max (a product of Q and the arterial content of oxygen (CaO2)) is also reduced because Q cannot increase above Qmax to compensate for decreased CaO2.

   When VO2max is reduced at altitude, metabolic rate at a given workload represents a higher relative intensity (i.e. percentage of VO2max). This increased intensity required for a certain workload is reflected in a reduced time to exhaustion at a constant work rate or an increased time to completion for constant task events. During submaximal exercise, when CaO2 is reduced, HR, ventilation, and Q are increased to maintain O2 delivery at a given intensity. The reduction in exercise economy is most notable in endurance events. According to Fulco et al, events lasting less than two minutes are essentially unaffected by altitude. Events greater than two minutes in duration see significant increases in race completion times.

   Hypoxia-induced pulmonary hypertension has also been associated with intra-pulmonary arteriovenous anastomoses (shunts). It has been hypothesized that shunts act as a release mechanism for increased PAP. In situations where pulmonary pressures are increased pathologically, the shunts open, allowing blood to bypass pulmonary circulation relieving pressure. It is also possible that shunts reduce the deleterious effect of right ventricular (RV) afterload on Q (caused by increased PAP), and allow an increase in Q. Several studies show that shunts are minimal to non-existent in most humans at rest, but both exercise and hypoxia are significant stimuli to cause shunt opening. Shunting appears to occur more frequently in some subjects in hypoxia while others remain unaffected.

   A strategy used to mitigate the performance decline at altitude is to lower PAP by promoting pulmonary arteriole smooth muscle relaxation pharmaceutically. Phosphodiesterase (PDE) inhibitors act on the nitric oxide (NO) system in smooth muscle to reduce pulmonary artery pressure. The mechanism and effect of the PDE inhibitor sildenafil will be examined as a performance enhancer in hypoxic exercise conditions.

   Originally investigated as an anti-angina medication, sildenafil has been successfully used to treat pulmonary arterial hypertension and erectile dysfunction because of its vasodilatory properties on the NO pathway. Sildenafil is a PDE-5 inhibitor with a similar molecular structure to cGMP. By competing with cGMP (cyclic guanosine monophosphate) for binding sites on PDE-5, sildenafil prevents cGMP breakdown, increasing the concentration available for smooth muscle relaxation. Sildenafil does not increase smooth muscle relaxation by increasing NO availability, but by inhibiting the mechanism that reduces the effects of NO.

   In addition to its therapeutic use, sildenafil has recently been studied for its potential to enhance exercise performance, specifically in hypoxia. Ghofrani et al. were the first to report the effects of sildenafil on exercise performance in hypoxia and found a significant improvement in exercise capacity. Ghofrani hypothesized that sildenafil would improve hypoxic exercise tolerance by blunting the pulmonary hypertensive response, decreasing PAP and thereby reducing RV afterload allowing an increase in Q.

   Subsequent studies have attempted to elucidate the mechanism through which sildenafil might improve performance with mixed success. Because increases in mean power output during a time-trial are directly related to performance outcomes, there is significant potential for sildenafil to be used as an ergogenic aid in endurance sport. Despite the logical rationale, the results of subsequent investigations into the ergogenic potential of sildenafil have been inconsistent, some show a benefit in hypoxia and others show no significant effect when compared to placebo.

   Sildenafil is an effective pulmonary vasodilator in hypoxia, and does increase Q. In the 2006 study by Hsu et al, several subjects showed a significant improvement in time-trial performance following sildenafil administration. These subjects also showed an exaggerated decline in exercise performance in hypoxia. By grouping their subjects according to those with a greater than or less than one minute improvement in time-trial performance between placebo and sildenafil, the authors classified subjects as responders and non-responders. The responders had higher pulmonary vascular resistance (PVR) due to increased PAP and resultant increased RV afterload. In these subjects, sildenafil improved performance by decreasing PAP and PVR, reducing RV afterload, and improving V/Q mismatch. Non-responders had no such increases in PAP, PVR, or performance after taking sildenafil. Kressler et al, acknowledge that responders as described by Hsu may represent only a small fraction of the population and may not have been included in the second study.

   The differences in responders and non-responders could be explained by the inter-individual variability in the HPV response. Some humans have a much more robust HPV response where pulmonary blood flow is dramatically reduced, causing significant decreases in PAP and Q. Others may have a nearly non-existent HPV response allowing blood flow to remain relatively unchanged even during hypoxic exercise. Similarly, there is high inter-individual variability in the exercise performance response to hypoxia. Some athletes perform poorly at altitude, while others performance is relatively unaffected. We believe that poor performance at altitude may be the result of a robust HPV response and that sildenafil may act to equalize this, bringing those with a robust HPV response to the same level as those with a minimal response.
4. Objectives

   The objective of the first phase of the study is to evaluate the HPV response in normoxia (with placebo), hypoxia (with placebo), and hypoxia (with sildenafil) using both steady-state exercise and a time-trial race simulation. Cardiopulmonary variables including pulse oxygen saturation (SPO2), heart rate (HR), ventilation, (VE), and oxygen consumption (VO2) will be measured. During steady-state exercise, PAP and cardiac output (Q) will be measured using the tricuspid jet method. During the time-trial, time to completion and average power will be recorded.

   The objective of the second phase of the study is to determine the magnitude of responses in HPV, HVR, and shunt in various levels of hypoxia and if this response is reduced with sildenafil.
5. Research Method

Participants: Ten healthy, male or female, competitive cyclists will be recruited to participate in the study. Participants will be recruited using advertisements posted on campus and distributed electronically to local cycling clubs. Participants must refrain from the consumption of alcohol or caffeine, foods high in nitrates including beets and green leafy vegetables, and abstain from vigorous exercise for 24 hours prior to each visit.

Familiarization: Subjects will report to the Environmental Physiology Laboratory (EPL) to sign informed consent and be familiarized with the metabolic cart and hypoxic chamber. This visit will take approximately 1 hour.

Pre-testing: Each subject will begin by completing a screening test including pulmonary function testing (PFT) using spirometry to measure forced expiratory volume in one second (FEV1) and forced vital capacity (FVC). Subjects will perform a baseline, ramp VO2max test using a stationary cycle ergometer and a metabolic cart. Work rate will start at 100 Watts (W), and increase by 30 W/min until volitional exhaustion. Expired gases will be collected in a mixing chamber to determine VO2max as an estimate of aerobic fitness. Fifteen minutes after completing the normoxic test, the subject will complete a second, hypoxic (FIO2 = 0.16) baseline ramp test. This visit will take approximately 1.5 hours. Following successful admittance to the study, a second session will be scheduled.

Study Sessions (Phase 1): Once admitted to the study, subjects will report to the EPL on three occasions for Phase 1 of the study, where they will complete one hypoxic (FIO2 = 0.16) practice and three (randomized) experimental (one hypoxic control: FIO2 = 0.16 with placebo, one hypoxic sildenafil: FIO2 = 0.16 with sildenafil, and one normoxic control: FIO2 = 0.21 with placebo) 15km time-trials. Each experimental trial will be separated by one week. One hour prior to the time-trial, subjects will be given either 50mg sildenafil or placebo. After an hour, a 4ml venous blood sample will be taken to test for serum sildenafil levels. Subjects will be asked to complete a self-selected warm-up on the cycle ergometer as if they are preparing for a race. Following warm-up, subjects will cycle for 15 minutes at a power output corresponding to 50% of their peak power (determined in pre-testing) in normoxia or hypoxia. Upon completion of the steady-state portion, subjects will be allowed to rest for 5 minutes before beginning their 15km time-trial. Throughout the exercise bout, expired gases will be collected using a metabolic cart to measure cardiopulmonary parameters (SPO2, HR, ventilation (VE) and VO2). During the steady-state portion, cardiac output will be measured with Doppler echocardiography. Pulmonary artery pressure will be estimated by echocardiography of the tricuspid jet performed by a trained sonographer. During time-trial exercise, performance variables (time to completion and mean power output) will be recorded. Each visit will take approximately 2.5 hours.

The experiment will utilize a randomized, double blind, crossover design. Participants will complete the entire protocol after sildenafil once and placebo twice and researchers will be blinded to the condition. A computerized random number generator will determine the order in which the trials are completed. In both normoxic and hypoxic conditions, the subject will breathe air supplied by the EPL hypoxic chamber. The chamber can be operated both at simulated altitude and sea-level. By setting the chamber to ambient air conditions, the subject is blinded to the condition as they are still breathing air from the chamber, which is on and making the same noise and at the same humidity as if simulating altitude.

Data Analysis: During steady-state and the time-trial, mean SPO2, HR, VE, VO2, Q and PAP during the final five minutes of the steady-state and the entire time trial will be compared using analysis of variance (ANOVA) between sea-level placebo, hypoxic placebo, and hypoxic sildenafil. The decrease in time-trial mean power output (Δ power) will be determined between hypoxia and normoxia with placebo and will be compared to the increase in mean PAP (Δ PAP) and decreased Q (Δ Q) by determining the correlation coefficient. Multivariate regression analysis will be used to compare the dependent variables (SPO2, VO2, PAP, and Q) with the effect of sildenafil on mean power output in hypoxia.

During steady-state exercise and time-trial in hypoxia, we expect to observe significant decreases in SPO2, VO2, and Q, and significant increases in HR, VE, and PAP compared to sea-level. We hypothesize that decreases in time-trial mean power output in hypoxia are the result of (and thus will be negatively correlated with) increases in pulmonary artery pressure and accompanied by a decrease in Q. We believe sildenafil will reduce PAP and increase Q, allowing an increase in mean power output.

Study Sessions (Phase 2): Subjects will report to the EPL and sildenafil (50 mg) or placebo will be administered (order of administration to be determined randomly by computer assignment). One hour after ingesting the pill, a 4ml venous blood sample will be taken. Subjects will be tested for intrapulmonary shunt and PAP will be measured during different levels of hypoxia (FIO2= 0.21, 0.16, 0.12) corresponding to sea-level, 2500 meters, and 4500 meters. Shunt will be determined using the agitated saline contrast echocardiography technique. Hypoxic gas will be generated using mixed O2 and N2 contained in a large mixing chamber and delivered to the subject via tubing and a one-way non-rebreathing mask. The procedure will be repeated with the remaining medication and no less than one week between trials. Each visit will take approximately two hours.

The experiment will utilize a randomized, double blind, crossover design. Participants will complete the entire protocol after taking sildenafil and placebo and researchers will be blinded to the condition. A computerized random number generator will determine the order in which the trials are completed. In both normoxic and hypoxic conditions, the subject will breathe air from a large mixing chamber (balloon).

Data Analysis: A 3x2 analysis of variance (ANOVA) will be used to compare the effects of hypoxia (sea-level, moderate hypoxia, and severe hypoxia) and medication (sildenafil and placebo) on SPO2, VE, VO2, Q, and PAP at rest. A 3x2x2 ANOVA will be used to assess the effects of hypoxia (sea-level, moderate hypoxia, and severe hypoxia), medication (sildenafil and placebo), and presence of intrapulmonary shunt (present or not present) on PAP.

At rest, with increasing levels of hypoxia we expect increases in VE, VO2, and PAP and decreases in SPO2, and Q. These changes will be reduced with sildenafil compared to placebo. At any given level of hypoxia, subjects with intrapulmonary shunts present will exhibit a higher PAP and lower SPO2. With sildenafil, fewer subjects will exhibit pulmonary shunting in hypoxia and PAP will be decreased.

ELIGIBILITY:
Inclusion Criteria:

* between age 19 (18 if a University of British Columbia student) and 40
* healthy
* competitive cyclist (hold current racing license of professional, category 1, or 2 or have a measured VO2max greater than 60 ml.min.kg).

Exclusion Criteria:

* smokers
* anyone unable to complete the exercise protocol
* individuals with a history of cardiovascular or respiratory illness
* those with an atrial or ventricular septal defect (e.g. patent foramen oval)
* anyone currently prescribed sildenafil, tadalafil, vardenafil or any other PDE-5 inhibiting medication
* anyone who has lived more than 15 days at moderate altitude in the last three months

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
Performance in completion of Time Trial task | 20 minutes after test.
  Performance is measured as the mean power output achieved during the time trial task.

SECONDARY OUTCOMES:
PAP measured with ultrasound during exercise. | 20 minutes after test.
  PAP is measured in mmHg at the tricuspid jet.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Carter, MSc, Study Director — UBC; Michael Koehle, MD, PhD, Principal Investigator — UBC
Locations (1):
- University of British Columbia - Environmental Physiology Laboratory, Vancouver, British Columbia, Canada